CLINICAL TRIAL: NCT03955510
Title: Abnormal Food Timing and Circadian Dyssynchrony in Alcohol Induced Colon Carcinogenesis
Acronym: AFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Professor, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 16051904
Record Dates: First submitted 2019-04-08; First posted 2019-05-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sigmoidoscopy; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "Right-time eating" / no alcohol (Other): "Right-time eating" means breakfast before 8am, lunch before 1 pm and dinner before 6pm. Subjects will be asked to stick to this eating schedule for 1 week. Subjects will be asked to not drink alcohol for 1 week. Subjects will randomly be assigned to each eating pattern during the study period.
  Interventions: Other: Right time eating; Procedure: Sigmoidoscopy; Procedure: Optional 24h circadian assessment in the Biological Rhythms lab
- "Right-time eating" / with alcohol (Other): "Right-time eating" means breakfast before 8am, lunch before 1 pm and dinner before 6pm. Subjects will be asked to stick to this eating schedule for 1 week. Subjects will randomly be assigned to each eating pattern during the study period. Moderate alcohol drinking means 0.3-0.5 g/kg alcohol daily, which will be not more than 2 glasses of wine depending on subject's weight. Alcohol will always be consumed in the evening with food or after food (e.g., dinner). The timing of alcohol consumption will be consistent for each individual. Subjects will be provided with red wine for the 1 alcohol intervention week. The order of conditions will be random.
  Interventions: Other: Right time eating; Procedure: Sigmoidoscopy; Procedure: Optional 24h circadian assessment in the Biological Rhythms lab; Other: Alcohol
- "Delayed-eating" / no alcohol (Other): "Delayed-eating" means eating each meal 3 hours later than the "Right-time eating."Subjects will be asked to stick to this eating schedule for 1 week. Subjects will randomly be assigned to each eating pattern during the study period. Subjects will be asked to not drink alcohol for 1 week.
  Interventions: Other: Delayed time eating; Procedure: Sigmoidoscopy; Procedure: Optional 24h circadian assessment in the Biological Rhythms lab
- "Delayed-eating" / with alcohol (Other): "Delayed-eating" means eating each meal 3 hours later than the "Right-time eating."Subjects will be asked to stick to this eating schedule for 1 week. Subjects will randomly be assigned to each eating pattern during the study period. Moderate alcohol drinking means 0.3-0.5 g/kg alcohol daily, which will be not more than 2 glasses of wine depending on subject's weight. Alcohol will always be consumed in the evening with food or after food (e.g., dinner). The timing of alcohol consumption will be consistent for each individual. Subjects will be provided with red wine for the 1 alcohol intervention week. The order of conditions will be random.
  Interventions: Other: Delayed time eating; Procedure: Sigmoidoscopy; Procedure: Optional 24h circadian assessment in the Biological Rhythms lab; Other: Alcohol

INTERVENTIONS:
Other: Right time eating — "Right-time eating" means breakfast before 8am, lunch before 1 pm and dinner before 6pm. Subjects will be asked to stick to this eating schedule for 1 week. Subjects will randomly be assigned to each eating pattern during the study period. Each subject will be required to do this intervention twice during the study period. One time they will have right time eating with alcohol , the second time the will have this intervention without alcohol.
  Arms: "Right-time eating" / no alcohol; "Right-time eating" / with alcohol
Other: Delayed time eating — "Delayed-eating" means eating each meal 3 hours later than the "Right-time eating."Subjects will be asked to stick to this eating schedule for 1 week. Subjects will randomly be assigned to each eating pattern during the study period. Each subject will be required to do this intervention twice during the study period. One time they will have delayed time eating with alcohol , the second time the will have this intervention without alcohol.
  Arms: "Delayed-eating" / no alcohol; "Delayed-eating" / with alcohol
Procedure: Sigmoidoscopy — Subjects will undergo unprepped sigmoidoscopy to collect tissue and stool sample at each intervention visits (visit 2, 3, 4, and 5). Flexible sigmoidoscopy will not require any colon cleansing and it will be very limited to the most distal (closest to the end of the anus) 20 centimeters (approximately 8 inches) of the colon and thus will be far less uncomfortable than the routine flexible sigmoidoscopy.
Procedure: Optional 24h circadian assessment in the Biological Rhythms lab — Subjects may choose to participate in the 24 hour circadian assessment in the Biological Rhythms Research Lab. During this assessment, a saliva sample will be taken every hour, a mouth swab will be done every 2 hours, and rectal swab will be done twice (every 12 hours). Subjects will be kept awake in dim light on a recliner chair. Subjects can watch a television with dimmed light. Subjects will be provided with food and drink during the assessment.
  If subjects choose this intervention they will be asked to complete 4 assessment during the course of the study period.
Other: Alcohol — Moderate alcohol drinking means 0.5 g/kg alcohol daily, which will be not more than 2 glasses of wine depending on subject's weight. Alcohol will always be consumed in the evening with food or after food (e.g., dinner). The timing of alcohol consumption will be consistent for each individual. Subjects will be provided with red wine for the 2 alcohol intervention weeks. The order of conditions will be random.
  Arms: "Delayed-eating" / with alcohol; "Right-time eating" / with alcohol

SUMMARY:
The purpose of this study is to study the impact of Western lifestyle, including moderate alcohol consumption and delayed eating patterns on studying individuals' susceptibility to colorectal cancer. This study aims to increase our ability to identify individuals at risk for colorectal cancer in the future.

Each subject will experience four conditions (each for one week in duration with a week +/- 2 days wash-out in between): (1) "right-time eating" / no alcohol, (2) "right-time eating" / with alcohol, (3) "delayed-eating" / no alcohol, (4) "delayed-eating" / with alcohol. The order of experiments will be randomized [concealed randomization]. All subjects will undergo unprepped sigmoidoscopy after each week of intervention. In Aim 2, all subjects will have an option to undergo a 24h circadian assessment in the Biological Rhythms Research Lab after each week of intervention. The Investigator will assess (i) central circadian rhythms by collecting hourly salivary samples for melatonin assays and (ii) peripheral rhythm in the intestinal tract by buccal swabs once every 2h (12 time points) as well as by rectal sampling twice (every 12 hr). For Aim 3, sigmoidoscopy without sedation will be used to obtain colonic samples as the safe method compared to colonoscopy, which has some small but finite risks associated with the procedure (e.g, bleeding or perforation) as well as sedation.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer mortality in the US. CRC's risk is closely linked to the modern lifestyle. Alcohol is commonly used in our society and is an established risk factor for both pre-cancerous (polyp) and cancerous lesions of the colon. However this knowledge has not been translated to our current risk stratifications for CRC as the process of alcohol-induced carcinogenesis is not predictable. Mucosal inflammation is a well-established mechanism that mediates the effect of alcohol induced tissue injury in the intestine. Inflammation also plays a crucial role in pathogenesis of CRC. Factors that promote a pro-tumorigenic inflammatory state in the setting of alcohol are unknown. Since CRC occurs only in a small subset of alcohol user, alcohol alone may not be sufficient to start the neoplastic process and additional cofactors are required. One such factor is circadian dysrhythmia that is another modern lifestyle habit, shown to be associated with an increased risk of CRC. Further, previous research has shown that disruption of circadian rhythm exacerbates alcohol-induced intestinal inflammation. The Investigator hypothesize that altered circadian rhythms due to "wrong-time" eating (abnormal eating) are an important determinant in alcohol induced mucosal inflammation and carcinogenesis. Our preliminary data supports our hypothesis and shows that abnormal eating patterns accelerate alcohol-induced polyposis in a mouse model of CRC. Each subject will experience four conditions (each for one week in duration with a week +/- 2 days wash-out in between): (1) "right-time eating" / no alcohol, (2) "right-time eating" / with alcohol, (3) "delayed-eating" / no alcohol, (4) "delayed-eating" / with alcohol. The order of experiments will be randomized [concealed randomization]. All subjects will undergo unprepped sigmoidoscopy after each week of intervention. In Aim 2, all subjects will have an option to undergo a 24h circadian assessment in the Biological Rhythms Research Lab after each week of intervention. The Investigator will assess (i) central circadian rhythms by collecting hourly salivary samples for melatonin assays and (ii) peripheral rhythm in the intestinal tract by buccal swabs once every 2h (12 time points) as well as by rectal sampling twice (every 12 hr). For Aim 3, sigmoidoscopy without sedation will be used to obtain colonic samples as the safe method compared to colonoscopy, which has some small but finite risks associated with the procedure (e.g, bleeding or perforation) as well as sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (greater than 21 years old)
2. Have had advanced tubular adenoma within the last year

Exclusion Criteria:

1. Asian ethnicity (Due to common polymorphisms of enzymes involved in alcohol metabolism)
2. Does not drink alcohol
3. Alcohol use disorder/Alcohol Abuse
4. A known genetic predisposition to colorectal cancer (FAP, Lynch syndrome)
5. A history of colorectal cancer or inflammatory bowel diseases
6. Presence of comorbidities that might affect the circadian system

   1. Chronic renal failure
   2. Cirrhosis
   3. Advanced neurological conditions (e.g., Parkinson's, MS, epilepsy)
   4. Psychological disorders (e.g., PTSD, major depression)
   5. Sleep apnea
   6. Restless Leg Syndrome
   7. Inpatient Status
   8. Advanced cardiac failure
   9. Night shift workers with active shift work in the past month
   10. Planned shift work that will occur during the study
   11. Crossed more than two time zones in the previous week
7. Conditions that alter or necessitate a particular eating pattern (e.g., uncontrolled diabetes, eating disorders)
8. Conditions that alter the microbiota (infection or recent history of antibiotic use within three months, or use of pro/prebiotics within one month prior to recruitment)
9. Regular use of medications that can potentially affect melatonin profiles (e.g., Melatonin, Metoclopramide, Psychotropic medications, Hypnotics during the four weeks prior to the study)
10. Any active cancer
11. Inability to sign an informed consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mucosal Outcome | Through study completion and data analysis in 3 years (2022)
  Sigmoid mucosal biopsy specimens are collected at baseline and at the end of each intervention week. Using gene expression analysis (RNA seq), impact of our intervention on sigmoid mucosal samples, with regard to the mucosal immune response will be assessed. This will be assessed by % change in immune expression.
  Tissue staining will be used to measure the effect of our interventions on markers of colonic neoplastic process including epithelial proliferation and apoptosis. The effect will be assessed by % changes in proliferation and apoptosis rate in the tissue.
Circadian Outcome | Through study completion and data analysis in 3 years (2022)
  Impact of our treatments on circadian read outs will be assessed by using a wrist actigraphy in which activity data to calculate phase assessment (hr units) and sleep indexes including {sleep duration, wake after sleep onset (in minutes), total sleep time (in minutes), and sleep percentage} will be measured.
  If the subject is interested, our in house circadian lab measurements (activity data and urine melatonin as described plus buccal circadian gene expression) will be available to complement the aforementioned circadian measures. To this end , subjects will enter the Biological Rhythms Research Lab after each week of the intervention period for 24h for assessments of central circadian rhythms (hourly salivary melatonin) and peripheral clock genes of the digestive tract from mucosal cells taken from buccal swaps once every 2h (12 time points). Percent change in expression level of the genes will be compared between groups.
Microbiota Outcome | Through study completion and data analysis in 3 years (2022)
  Microbial DNA will be isolated from the stool and the biopsy material Effects of the interventions in this study on the gut microbial compositions will be identified by using 16s microbial analysis.

SECONDARY OUTCOMES:
Food time and Sleep time Outcomes | Through study completion and data analysis in 3 years (2022)
  Eating and sleeping time will be recorded by having participants complete the weekly Food Timing/Sleep Questionnaire where participants record their meal timings and sleep hours throughout the period of the study. Variation in meal and sleep time in weekdays and weekends (in hour unit) will be compared among conditions.
Gastrointestinal symptoms | Through study completion and data analysis in 3 years (2022)
  Subjects may report their experience after each intervention. For this, we will provide participants a questionnaire about common gastrointestinal symptoms that they have experienced within the past 7 days. Participants will scale the severity of their symptoms from 0 - 10 (1 being very mild, 10 being very severe and 0 if no symptom experienced).
A 24h food recall | Through study completion and data analysis in 3 years (2022)
  24h food recall will be completed by participants using Automated Self-Administered 24-Hour at baseline and once during each intervention.
Establish the link and interaction of delayed eating, and alcohol intake on risks associated with colon cancer. | Through study completion and data analysis in 3 years (2022)
  Effects of delayed eating with alcohol on circadian outcome, microbiota and mucosal markers of colon carcinogenesis will be assessed by analyzing neoplastic mucosal markers (via tissue staining) as well as gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No identifying information will be shared with other researchers

DOCUMENTS (2):
  • Study Protocol: AFT with cover page (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03955510/Prot_000.pdf
  • Informed Consent Form (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03955510/ICF_001.pdf